CLINICAL TRIAL: NCT03318497
Title: Initial Evaluation of Role of Early Interim 18F-FLT PET/CT for Outcome Prediction in Pancreatic Adenocarcinoma
Brief Title: Role of Interim 18F-FLT PET/CT for Outcome Prediction in Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Daniella Pinho, Assistant Professor, Radiology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 012017-029 Protocol V6
Record Dates: First submitted 2017-10-06; First posted 2017-10-24 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; 18F-FLT; FLT; Locally advanced pancreatic adenocarcinoma; Borderline resectable pancreatic adenocarcinoma; resectable pancreatic adenocarcinoma
MeSH Terms: interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: The interim 18F FLT-PET/CT will be performed after the 2nd cycle of chemotherapy regimen, but before the commencement of 3rd cycle.
  Clinical Follow Up: Standard of care clinical follow-up data will be collected up to 2 years following the end of chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Interim FLT PET/CT) (Experimental): The experimental 18F-FLT-PET/CT is required to be completed before initiation of chemotherapy. Labs and correlative radiology, as directed per clinical care, are required within 30 days prior to 18F-FLT-PET/CT; and 18F-FDG-PET/CT is required within 30 days before the 18F-FLT-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.
  * Procedure: Computed Tomography
  * Drug: 3'-deoxy-3'-[F-18] fluorothymidine: [F-18]FLT
  * Other: Laboratory Biomarker Analysis
  * Procedure: Positron Emission Tomography
  Interventions: Drug: 3'-deoxy-3'-[F-18] fluorothymidine: [F-18]FLT; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: 3'-deoxy-3'-[F-18] fluorothymidine: [F-18]FLT — Given IV The experimental 18F-FLT-PET/CT is required to be completed before initiation of chemotherapy. Labs and correlative radiology, as directed per clinical care, are required within 30 days prior to 18F-FLT-PET/CT; and 18F-FDG-PET/CT is required within 30 days before the 18F-FLT-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.
  Other Names: FLT; 3'-deoxy-3'-[F-18] fluorothymidine
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT SCAN
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
To assess if percentage change in 18F-FLT PET/CT quantitative parameters (SUV max, or SUV peak or proliferative tumor volume) after 2 cycles of neoadjuvant chemotherapy can predict overall survival at 1 and 2 years and progression free survival at 6 months and 1 year in patients with borderline resectable or locally advanced, pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The experimental 18F-FLT-PET/CT is required to be completed before initiation of chemotherapy. Labs and correlative radiology, as directed per clinical care, are required within 30 days prior to 18F-FLT-PET/CT; and 18F-FDG-PET/CT is required within 30 days before the 18F-FLT-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.

Visit 1: Patients will have at least one visit with investigator (or investigator designee) prior to the study to review clinical history and prior treatment of pancreatic adenocarcinoma, and to explain the study. Correlative radiology studies including CT, MRI and 18F FDG-PET/CT as per institutional routine clinical care, and any clinically-directed laboratory tests performed as part of staging must be performed within 30 days of the 18F FLT-PET/CT

Visit 2 (Optional): The 18F-FDG-PET/CT may be done as a research scan, if the patient is unable to obtain a clinically-directed 18F-FDG-PET/CT as part of their clinical care or within 30 days of 18F FLT-PET/CT. The research 18F-FDG-PET/CT, in this instance, will be identical in procedure to the institution's clinical 18F-FDG-PET/CT. The blood glucose level will be < 200 mg/dl, before 18F-FDG injection, which is institutional standard clinical protocol. The following additional patient data will be obtained: histological diagnosis of primary and/or metastatic disease, date of diagnosis of primary and metastatic disease, gender, height, weight (for BMI), ECOG score and confirmation of absence of prior treatment.

Visit 3: Day of 18F-FLT-PET/CT: The patient will have an intravenous line placed in the hand or arm, 18F-FLT-PET/CT will be given by 1-2 minute IV push, and the dose administered will be approximately 5 mCi (+/- 20% dose). After approximately 60 +/- 10 minutes of uptake time, the patient will be positioned supine in the PET/CT scanner for standard whole body PET/CT scan from the skull base to mid-thigh. This scan will take approximately 20-30 min. The window from FLT PET/CT baseline study to initiation of chemotherapy should be no more than 30 days.

Visit 4: Day of Interim 18F-FLT-PET/CT: The interim 18F FLT-PET/CT will be performed after the 2nd cycle of chemotherapy regimen, but before the commencement of 3rd cycle. The second 18F-FLT-PET/CT study must be performed on the same scanner as the first 18F FLT-PET/CT and the imaging protocol described in Visit 3 should be closely followed.

Study duration:

Clinical Follow Up: Standard of care clinical follow-up data will be collected up to 2 years following the end of chemotherapy.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed pancreatic adenocarcinoma (resectable, borderline resectable or locally advanced disease at presentation) are eligible for the study.
* Patients should not have any type of curative or palliative therapy for pancreatic adenocarcinoma before enrolling in the study.
* Patients must be over 18 years old and capable and willing to provide informed consent.
* Patients must have measurable disease (by RECIST 1.1 criteria)
* Patients must have an ECOG performance status of 0-3 (restricted to ECOG PS 0-2 if age >70 years).
* Patients of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to FLT (or FDG if for research) PET/CT imaging per institution's standard of care; A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria; Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Medically stable as judged by patient's physician.
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals of similar chemical or biologic composition to FLT are NOT eligible.
* Ability to understand and the willingness to sign a written informed consent.
* Patient must be able to lie still for a 20 to 30 minute PET/CT scan.

Exclusion Criteria:

* Subjects who had prior chemotherapy or radiotherapy for pancreatic adenocarcinoma cannot participate in the study.
* Patient must NOT be pregnant or breast-feeding.
* Patients have no clinical evidence of distant metastatic disease
* Patients must not weigh more than the maximum weight limit for the table for the PET/CT scanner where the study is being performed.(>200kg or 440lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Pinho, MD, Principal Investigator — UT Soutwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Interim FLT PET/CT): The experimental 18F-FLT-PET/CT is required to be completed before initiation of chemotherapy. Labs and correlative radiology, as directed per clinical care, are required within 30 days prior to 18F-FLT-PET/CT; and 18F-FDG-PET/CT is required within 30 days before the 18F-FLT-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.
  * Procedure: Computed Tomography
  * Drug: 3'-deoxy-3'-[F-18] fluorothymidine: [F-18]FLT
  * Other: Laboratory Biomarker Analysis
  * Procedure: Positron Emission Tomography
    3'-deoxy-3'-[F-18] fluorothymidine: [F-18]FLT: Given IV The experimental 18F-FLT-PET/CT is required to be completed before initiation of chemotherapy. Labs and correlative radiology, as directed per clinical care, are required within 30 days prior to 18F-FLT-PET/CT; and 18F-FDG-PET/CT is required within 30 days before the 18F-FLT-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.
  Computed Tomography: Undergo PET/CT
  Positron Emission Tomography: Undergo PET/CT
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Diagnostic (Interim FLT PET/CT)
Started | 6
Completed | 2
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Summed Standardized Uptake Value (SUVmax) of Lesion After 2 Cycles of Chemotherapy
Description: Change in FLT PET/CT SUV Max after 2 cycles of chemotherapy will be compared to baseline (pre-treatment FLT PET/CT SUV Max)
Time Frame: Baseline(pre-treatment), 2 cycles after starting chemotherapy (each cycle 14 days)
Population: Only two of the enrolled subjects completed both 18F-FLT-PET/CT scans.
Measure: Mean (Full Range); unit: percentage of SUV Max change
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 2
percentage of SUV Max change | 27.45 [-35.8 to 90.96]

2. Primary Outcome: Change From Baseline in SUV Peak of Lesion After 2 Cycles of Chemotherapy
Description: Change in FLT PET/CT SUV peak after 2 cycles of chemotherapy will be compared to baseline (pre-treatment FLT PET/CT SUV Peak)
Time Frame: Baseline(pre-treatment), 2 cycles after starting chemotherapy (each cycle 14 days)
Population: Data was not collected.
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 0

3. Primary Outcome: Change From Baseline in Proliferative Tumor Volume After 2 Cycles Chemotherapy
Description: Change in FLT PET/CT Proliferative tumor volume after 2 cycles of chemotherapy (compared to pre-treatment FLT PET/CT proliferative tumor volume)
Time Frame: Baseline(pre-treatment), 2 cycles after starting chemotherapy (each cycle 14 days)
Population: Data was not collected
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 0

4. Primary Outcome: 1 Year Overall Survival
Description: Proportion of subjects who were alive at 1 year post-treatment is assessed
Time Frame: Baseline(pre-treatment), until date of first observed death, assessed up to 1 year
Measure: Number; unit: percentage of subjects
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 6
percentage of subjects | 67

5. Primary Outcome: 2 Year Overall Survival
Description: Proportion of subjects who were alive at 2 years post-treatment is assessed
Time Frame: Baseline(pre-treatment), until date of first observed death, assessed up to 2 years
Measure: Number; unit: percentage of subjects
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 6
percentage of subjects | 33

6. Secondary Outcome: 6 Months Progression Free Survival
Description: Proportion of subjects who are progression free at 6 months post-treatment is assessed.
Time Frame: Baseline (pre-treatment), until date of first observed progression, assessed up to 6 months
Population: 1 subject died and data is not available to be reported
Measure: Number; unit: percentage of subjects
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 5
percentage of subjects | 40

7. Secondary Outcome: 1 Year Progression Free Survival
Description: Proportion of subjects who are progression free at 1 year post-treatment is assessed.
Time Frame: Baseline(pre-treatment), until date of first observed progression, assessed up to 1 year
Population: 1 subject died and data is not available to be reported
Measure: Number; unit: percentage of subjects
Arm/Group | Diagnostic (Interim FLT PET/CT)
Number analyzed (Participants) | 5
percentage of subjects | 40

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events after injection of the investigational agent and were contacted 24 hours after completion of PET/CT imaging to assess any potentially related adverse events. Subjects' medical records were monitored on a monthly basis to check for any additional adverse events, up 2 years.
Arm/Group | Diagnostic (Interim FLT PET/CT)
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03318497/Prot_SAP_004.pdf
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT03318497/ICF_003.pdf